CLINICAL TRIAL: NCT03868826
Title: Pain, Function and Quality of Life Before and After Treatment of Hamstring Avulsion
Status: Completed | Type: Observational
Sponsor: Horsens Hospital (Other)
Responsible Party: Principal Investigator, Jeppe Lange, Medical Doctor, PhD, Horsens Hospital
Other Study IDs: 1-16-02-75-19
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hamstring Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Orthopaedic surgery and/or rehabilitation — The avulsion is repaired and hereafter the patient follows rehabilitation. Some are treated conservatively and only follow rehabilitation.

SUMMARY:
The aim of the study is to investigate pain, function and quality of life before and 10-12 months after surgical repair and/or rehabilitation of hamstrings avulsion

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for treatment of hamstring avulsion

Exclusion Criteria:

* Conditions that contraindicate muscle strength testing e.g. cancer and neurological conditions
* Patients that do not speak or understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hamstring avulsion
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
Perth Hamstring Assessment Tool (PHAT) (0-100 scale) | Change from before surgery to 10-12 months after surgery on the 0-100 scale.
  Overall tool and pain subscale during sitting, steps and relaxing separately extracted. 0 indicates total problems and 100 no problems.
Knee flexion strength of affected leg (Newton meters per kilogram) | Change from before surgery to 10-12 months after surgery
  Maximal knee flexion strength of affected leg expressed as newton meters per kilogram, measured with a handheld dynamometer
Hip extension strength of affected leg (Newton meters per kilogram) | Change from before surgery to 10-12 months after surgery
  Maximal hip extension strength of affected leg expressed as newton meters per kilogram, measured with a handheld dynamometer
Overall health | Change from before surgery to 10-12 months after surgery on the 0-100 scale
  0-100 continuous scale (0 worst imaginable health, 100 best imaginable health)

SECONDARY OUTCOMES:
Knee flexion strength of contralateral leg (Newton meters per kilogram) | Change from before surgery to 10-12 months after surgery
  Maximal knee flexion strength of contralateral leg expressed as newton meters per kilogram, measured with a handheld dynamometer
Hip extension strength of contralateral leg (Newton meters per kilogram) | Change from before surgery to 10-12 months after surgery
  Maximal hip extension strength of contralateral leg expressed as newton meters per kilogram, measured with a handheld dynamometer
Hip Sports Activity Scale (0-8 scale) | Change from before surgery to 10-12 months after surgery on the 0-8 scale
  Type of activity before injury and present 0, no activity, 8 athlete level.

CONTACTS AND LOCATIONS:
Locations (1):
- Signe Kierkegaard, Horsens, Danmark, Denmark

REFERENCES:
- [Result] Spoorendonk K, Bohn MB, Storm JO, Lund B, Kierkegaard-Brochner S. Proximal Hamstring Avulsions: Surgical Versus Conservative Treatment Using a Shared Decision-Making Strategy. Orthop J Sports Med. 2024 Oct 21;12(10):23259671241275656. doi: 10.1177/23259671241275656. eCollection 2024 Oct. PMID 39440155